CLINICAL TRIAL: NCT02494635
Title: Ultrasound and Biomarker Tests of Bladder Cancer Invasiveness
Brief Title: Ultrasound and Biomarker Tests in Predicting Cancer Aggressiveness in Tissue Samples of Patients With Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: The PI left institution
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4B-15-5; NCI-2015-00862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-15-00245; 4B-15-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); P41EB002182 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-07-10 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Bladder Papillary Urothelial Carcinoma; Stage 0a Bladder Urothelial Carcinoma; Stage 0is Bladder Urothelial Carcinoma; Stage I Bladder Cancer With Carcinoma In Situ; Stage I Bladder Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma; Stage III Bladder Urothelial Carcinoma; Stage IV Bladder Urothelial Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, bladder washings, and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic (ultrasound, biomarker studies): Previously collected tumor tissue samples, bladder washings, and urine cells are stained with calcium dye, washed and immersed in external buffer solution, and then transferred to the ultrasound imaging system. Tissue, bladder wash cells and urine cells samples are also analyzed for biomarkers of invasiveness derived from or related to REST gene via qRT-PCR, Western blot, and FISH.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Biomarker analysis

SUMMARY:
This research trial studies two types of tests, an ultrasound test and a biomarker test, to see how well they predict how aggressive (invasive) bladder cancer is in samples from patients with bladder cancer. The aggressiveness of a tumor means how likely it is to invade the body and spread. The ultrasound test uses a fluorescent dye and stimulates cells under a microscope to see how they respond. This may allow doctors to predict how likely the cancer cells are to spread in the body. The biomarker test uses laboratory testing of samples from patients to study genes and other molecules that may predict the cancer invasiveness. Comparing two different ways of predicting cancer aggressiveness may help doctors identify how well they work, and may eventually allow doctors to predict aggressiveness without needing to take a biopsy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish an association between bladder cancer disease stage and the level of invasiveness as measured by a novel ultrasound assay.

II. To establish an association between bladder cancer disease stage and expression of novel invasiveness biomarkers related to the RE1-silencing transcription factor (REST) gene.

OUTLINE:

Previously collected tumor tissue samples, bladder washings, and urine cells are stained with calcium dye, washed and immersed in external buffer solution, and then transferred to the ultrasound imaging system. Tissue, bladder wash cells and urine cells samples are also analyzed for biomarkers of invasiveness derived from or related to REST gene via quantitative reverse transcriptase polymerase chain reaction (qRT-PCR), Western blot, and fluorescence in situ hybridization (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of UCC, having one of the stages (Ta, Tis, T1, and T2 or higher)
* Patients with UCC who are undergoing a standard procedure to remove cells/tissue from their bladders (cystoscopy, biopsy, or surgery)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the USC/Norris Comprehensive Cancer Center facilities with bladder cancer will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Observed change in fluorescence of responding cells using the cell response index (CRI) | Baseline to up to 30 minutes
  Data will be post-processed to determine the level of ultrasound-induced calcium response at each stimulus amplitude. Cell locations will be identified with CellProfiler image analysis software and used to extract the raw fluorescence intensities for each cell. CRI will be plotted against stimulus amplitude, a sigmoid will be fit to the curve, and threshold will be defined as the amplitude that yielded a 50% response.
Observed change in percentage of responding cells using the cell response index (CRI) | Baseline to up to 30 minutes
  Data will be post-processed to determine the level of ultrasound-induced calcium response at each stimulus amplitude. Cell locations will be identified with CellProfiler image analysis software and used to extract the raw fluorescence intensities for each cell. CRI will be plotted against stimulus amplitude, a sigmoid will be fit to the curve, and threshold will be defined as the amplitude that yielded a 50% response.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Weitz, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States